CLINICAL TRIAL: NCT06942039
Title: A Pilot Study of Intrathecal Topotecan and Maintenance Chemotherapy in the Post-consolidation Setting for the Treatment of High-risk Embryonal Central Nervous System Tumours in Children Less Than 6 Years of Age
Brief Title: Pilot Study of IT Topotecan and Maintenance Chemotherapy for HR-EBTs in Children < 6 Years, Post Consolidation
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: C17 Council (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DECRYPT-BABYBRAIN
Record Dates: First submitted 2025-04-09; First posted 2025-04-24 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-10

CONDITIONS: CNS Embryonal Tumor; CNS, Medulloblastoma; Atypical Teratoid Rhabdoid Tumor; Medulloblastoma, Childhood; Medulloblastoma, Group 3; Medulloblastoma, Group 4; Pineoblastoma; Neuroblastoma; Embryonal Tumor With Multilayered Rosettes; Embryonal Tumor With Abundant Neuropil and True Rosettes; Ependymoblastoma; Medulloepithelioma; CNS Embryonal Tumor With Rhabdoid Features; CNS Embryonal Tumor, Nos
Keywords: HR-EBT
MeSH Terms: conditions — Medulloblastoma; Rhabdoid Tumor; Pinealoma; Neuroblastoma; Neuroectodermal Tumors, Primitive; Pyloric Stenosis, Hypertrophic | interventions — Hydrocortisone; Cisplatin; Vincristine; Etoposide; Cyclophosphamide; Mesna; Filgrastim; Granulocyte Colony-Stimulating Factor; Carboplatin; Thiotepa; Tamoxifen; Isotretinoin; Celecoxib; etoposide phosphate; Temozolomide

STUDY DESIGN:
Intervention Model Description: All patients will receive 3 cycles of induction with IT chemotherapy and 3 cycles of consolidation therapy. Patients will then receive either Maintenance A or Maintenance B based on their risk profile.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comprehensive Multimodal Therapy Including Induction, Consolidation, and Risk-Adapted Maintenance (Experimental): Participants will undergo a comprehensive treatment regimen beginning with three 21-day cycles of Induction chemotherapy including intrathecal (IT) cytarabine with hydrocortisone, cyclophosphamide, etoposide, vinCRIStine, and cisplatin. Peripheral blood stem cells will be collected during this phase for later use. Patients who achieve complete response (CR) proceed directly to Consolidation; those who do not may undergo second-look surgery or national tumor board review.
  Consolidation consists of three 28-day cycles of CARBOplatin and thiotepa followed by autologous stem cell rescue. Patients then proceed to up to 48-54 weeks of Maintenance chemotherapy based on risk stratification.
  Low-risk patients receive monthly IT topotecan and a 28-day metronomic regimen including tamoxifen and ISOtretinoin.
  High-risk patients receive monthly IT topotecan and a more intensive regimen every 9 weeks including ISOtretinoin, celecoxib, etoposide, cyclophosphamide, and temozolomide.
  Interventions: Drug: Cytarabine IT; Drug: hydrocortisone; Drug: Cisplatin; Drug: Vincristine; Drug: Etoposide; Drug: Cyclophosphamide; Drug: Mesna; Drug: Filgrastim; Drug: carboplatin; Drug: Thiotepa; Drug: Topotecan IT; Drug: Tamoxifen; Drug: ISOtretinoin; Drug: Celecoxib; Drug: etoposide phosphate; Drug: Temozolomide

INTERVENTIONS:
Drug: Cytarabine IT — Age-based dosing as a part of double IT therapy (cytarabine, hydrocortisone) during induction (3 cycles, 1 cycle = 21 days) alongside CISplatin, vinCRIStine, etoposide, cyclophosphamide, mesna and filgrastim (G-CSF).
Drug: hydrocortisone — Double IT therapy (cytarabine, hydrocortisone) during induction (3 cycles, 1 cycle = 21 days) alongside CISplatin, vinCRIStine, etoposide, cyclophosphamide, mesna and filgrastim (G-CSF).
Drug: Cisplatin — Intravenous CISplatin given on Day 1 during induction (3 cycles, 1 cycle = 21 days) alongside double IT therapy, vinCRIStine, etoposide, cyclophosphamide, mesna and filgrastim (G-CSF).
  Other Names: CDDP
Drug: Vincristine — Intravenous VinCRIStine given on Days 1, 8 & 15 during induction (3 cycles, 1 cycle = 21 days) alongside double IT therapy, CISplatin, etoposide, cyclophosphamide, mesna and filgrastim (G-CSF).
  Other Names: VCR
Drug: Etoposide — Induction: Intravenous Etoposide given on Days 1, 2 & 3 during induction (3 cycles, 1 cycle = 21 days) alongside double IT therapy, CISplatin, vinCRIStine, cyclophosphamide, mesna and filgrastim (G-CSF).
  Maintenance Arm B (for high-risk patients): Oral Etoposide given on Days 1-21 every 9 weeks (max 6 cycles, 1 cycle = 9 weeks) in combination with IT Topotecan, ISOtretinoin, Celecoxib, Cyclophosphamide and Temozolomide.
Drug: Cyclophosphamide — Induction: Intravenous high-dose Cyclophosphamide given on Days 2 & 3 during induction (3 cycles, 1 cycle = 21 days) alongside double IT therapy, CISplatin, vinCRIStine, etoposide, mesna and filgrastim (G-CSF).
  Maintenance Arm B (for high-risk patients): Oral Cyclophosphamide given on Days 1-21 every 9 weeks (max 6 cycles, 1 cycle = 9 weeks) in combination with IT Topotecan, ISOtretinoin, Celecoxib, Etoposide and Temozolomide.
  Other Names: CPM
Drug: Mesna — Induction: Intravenous Mesna given at hour 0 of Cyclophosphamide delivery and 3, 6, 9 & 12 hours post-dose during induction (3 cycles, 1 cycle = 21 days).
Drug: Filgrastim — Induction: Subcutaneous or intravenous Filgrastim (G-CSF) given 24-48 hrs after last dose of chemotherapy and/or as per institutional guidelines until count recovery.
  Consolidation: Subcutaneous or intravenous Filgrastim (G-CSF) given 24-48 hours after last stem cell infusion and/or per institutional guidelienes until count recovery.
  Other Names: G-CSF
Drug: carboplatin — Consolidation: Intravenous Carboplatin given on days -3 & -2 during consolidation alongside thiotepa and filgrastim.
  Other Names: CARBO
Drug: Thiotepa — Consolidation: Intravenous Thiotepa given on days -3 & -2 during consolidation alongside carboplatin and filgrastim.
  Other Names: THIO
Drug: Topotecan IT — Maintenance A (for low-risk patients): IT Topotecan on Day 1 of each cycle (max 12 cycles, 1 cycle = 28 days) alongside Tamoxifen and ISOtretinoin.
  Maintenance B (for high-risk patients): IT Topotecan every 4 weeks (max 6 cycles, 1 cycle = 9 weeks) alongside ISOtretinoin, Celecoxib, Etoposide, Cyclophosphamide and Temozolomide.
  Other Names: Intrathecal Topotecan
Drug: Tamoxifen — Maintenance A (for low-risk patients): Oral Tamoxifen twice daily, Days 1-28 (max 12 cycles, 1 cycle = 28 days) alongside ISOtretinoin and IT Topotecan.
Drug: ISOtretinoin — Maintenance A (for low-risk patients): Oral ISOtretinoin twice daily on Days 15-28 of each cycle (max 12 cycles, 1 cycle = 28 days) alongside Tamoxifen and IT Topotecan.
  Maintenance B (for high-risk patients): Oral ISOtretinoin twice daily on Days 1-21, every 6 weeks (max 6 cycles, 1 cycle = 9 weeks) alongside IT Topotecan, Celecoxib, Etoposide, Cyclophosphamide and Temozolomide.
Drug: Celecoxib — Maintenance B (for high-risk patients): Oral Celecoxib twice daily on Days 1-21, every 6 weeks (max 6 cycles, 1 cycle = 9 weeks) alongside IT Topotecan, ISOtretinoin, Etoposide, Cyclophosphamide and Temozolomide.
Drug: etoposide phosphate — During Induction and Maintenance B (for high-risk patients), etoposide phosphate may be given for subsequent doses to patients who have experienced etoposide allergic reactions.
  Other Names: Etopophos
Drug: Temozolomide — Maintenance B (for high-risk patients): Oral Temozolomide daily on Days 1-21, every 9 weeks (max 6 cycles, 1 cycle = 9 weeks) alongside IT Topotecan, ISOtretinoin, Etoposide, Cyclophosphamide and Celecoxib.
  Other Names: TMZ

SUMMARY:
Pilot study to determine feasibility of adding intrathecal chemotherapy and maintenance therapy after high dose chemotherapy for treatment of newly diagnosed HR-EBTs in patients less than 6 years of age.

DETAILED DESCRIPTION:
This is a pilot study to determine feasibility of adding intrathecal (IT) chemotherapy and maintenance therapy after high dose chemotherapy for treatment of newly diagnosed HR-EBTs in patients less than 6 years of age. Patients meeting all inclusion criteria will receive 3 cycles of multiagent chemotherapy induction (vinCRIStine, cyclophosphamide, CISplatin, etoposide) with IT cytarabine and hydrocortisone, and 3 cycles of consolidation with CARBOplatin, thiotepa, and autologous stem cell rescue (as per CCG 99703). Maintenance chemotherapy will then be given immediately after the completion of consolidation therapy and consist of risk-stratified oral chemotherapy using either "Maintenance A" (48 weeks) using tamoxifen and retinoic acid or "Maintenance B" (54 weeks) using metronomic isotretinoin, celecoxib, etoposide, temozolomide, and cyclophosphamide. Both arms of maintenance will receive monthly IT topotecan.

Following the end of treatment, patients will be scheduled for a follow-up visit every 3 months for 24 months to evaluate PFS and OS. Approximately 15 patients will be recruited as part of this clinical study.

Patients aged between 0 and 6 years old at the time of enrollment will be eligible. This study will only enrol patients with high risk Central Nervous System Embryonal Brain Tumors (CNS-EBTs) with histologic and/or molecular confirmation of diagnosis for ATRT intrinsic to the brain and spinal cord, group 3 and group 4 MB, pineoblastoma, CNS neuroblastoma, ETMR, including embryonal tumor with abundant neuropil and true rosettes (ETANTR), ependymoblastoma and ETMR not otherwise specified), medulloepithelioma, CNS embryonal tumor with rhabdoid features (INI-1 intact) and CNS embryonal tumor, not otherwise specified.

Response to treatment will be evaluated using the modified RAPNO (Response Assessment in Pediatric Neuro-Oncology) 1.

This study will also explore the genetic landscape of CNS HR-EBTs. Our biological study will include genomic analyses of tumor and CSF with use of epigenomic analyses (methylation profiling) arrays, Nanostring sub-typing studies, Next generation sequencing analyses for DNA and/or RNA.

ELIGIBILITY:
Inclusion Criteria:

1. Tumor Tissue Sample
2. Age: Patient must be aged ≥ 0 years to ≤ 6 years at the time of definitive confirmation of histologic diagnosis of eligible CNS tumor.
3. Diagnoses. Participants must have Central nervous system (CNS) HR-EBT including atypical teratoid rhabdoid tumour (ATRT), group 3 and group 4 medulloblastoma (MB), pineoblastoma, CNS neuroblastoma, embryonal tumor with multi-layered rosettes (ETMR including embryonal tumor with abundant neuropil and true rosettes (ETANTR), ependymoblastoma and ETMR not otherwise specified), medulloepithelioma, CNS embryonal tumor with rhabdoid features (INI-1 intact) and CNS embryonal tumor, not otherwise specified. Metastatic disease included. Any extent of resection included.
4. Cranial and Spine MRI. A baseline MRI brain and spine with and without contrast is required for all patients. cranial MRI (with and without gadolinium) must be done pre-operatively. Post-operatively, cranial MRI (with and without gadolinium) must be done.
5. Lumbar Puncture (LP) CSF for cytopathology (strongly recommended but not mandatory; if medically feasible). A baseline LP CSF cytology either pre-operatively or post-operatively at least 10 days after definitive surgery for all patients if medically feasible (This is not mandatory and will not make the patient ineligible).
6. Life expectancy: Patients must have a life expectancy of greater than 8 weeks from diagnosis.
7. Performance level: Patients must have a performance status corresponding of a Lansky score ≥ 50.
8. Organ Function Requirements: Participants must have normal organ and marrow function as defined below:

Adequate renal function defined as:

- Creatinine clearance (12-24-hour urine collection) or radioisotope glomerular filtration rate (GFR) ≥ 60 ml/min/1.73m2

Adequate cardiac function defined as:

* Shortening fraction of ≥ 27% by echocardiogram, or
* Ejection fraction of ≥ 47% by radionuclide angiogram.

Adequate pulmonary function defined as:

- No evidence of dyspnea at rest and a pulse oximetry > 94% on room air.

Adequate Bone Marrow Function defined as:

* Peripheral absolute neutrophil count (ANC) > 1000/μL
* Platelet Count > 100,000/μL (without transfusion for 3 days)
* Hemoglobin greater than 8 gm/dL (may have received red blood cell (RBC) transfusions)

Adequate liver function defined as:

* Total bilirubin ≤ 1.5X upper limit of normal (ULN) within normal institutional limits for age (patients with documented Gilbert's Disease may be enrolled with Study Chair approval and total bilirubin ≤ 2.0 × ULN)
* Alanine Aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 100 U/L

Exclusion criteria:

1. Patients who are receiving any other conventional anti-cancer agents or investigational agents.
2. Patients who received previous therapy including radiotherapy or chemotherapy other than corticosteroids.
3. Presence of another malignancy, except if the other primary malignancy is neither currently clinically significant nor requiring active intervention.
4. Concomitant medications restrictions: Concurrent use of enzyme inducing anticonvulsants (e.g. phenytoin, phenobarbital, and carbamazepine), selected strong inhibitors of cytochrome P450 3A4 include azole antifungals, such as fluconazole, voriconazole, itraconazole, ketoconazole, and strong inducers include drugs such as rifampin, phenytoin, phenobarbitol, carbamazepine, and St. John's wort or CYP450 3A4 stimulators or inhibitors.
5. Other uncontrollable medical disease: Patient has a severe and uncontrollable medical disease (i.e., uncontrolled diabetes, hyperglycemia, chronic renal disease or active uncontrolled infection), has chronic liver disease (i.e., chronic active hepatitis and cirrhosis), hypercholesterolemia (serum cholesterol >300 mg/dL), intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, active hyperparathyroidism, or psychiatric illness/social situations that would limit compliance with study requirements.
6. Patients who have a known diagnosis of human immunodeficiency virus (HIV) infection, hepatitis B or C.
7. Ineligible diagnoses for study entry by neuropathology: This includes sonic hedgehog (SHH) and wingless (WNT) MBs, all ependymomas, all choroid plexus carcinomas, all high grade glial and glio-neuronal tumors, all diffuse midline gliomas, all primary CNS germ cell tumors, all primary CNS sarcomas, all primary or metastatic CNS lymphomas and solid leukemic lesions (chloromas, granulocytic sarcomas).
8. The participant or parent(s)/guardian(s) cannot comply with the study visit schedule and other protocol requirements, in the investigator's opinion.

All patients must meet inclusion/exclusion criteria prior to starting any protocol therapy.

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine the feasibility of adding intrathecal (IT) topotecan and maintenance therapy after high dose chemotherapy for treatment of newly diagnosed HR-EBTs in patients less than 6 years of age. | At completion of maintenance therapy (approximately 48-54 weeks after start of maintenance therapy)
  Feasibility failure will be defined by ≥5 patients who stop maintenance therapy (all IT and oral agents) due to excessive toxicity, deemed attributable to maintenance therapy
To test the feasibility of centralized diagnostics and national tumour board review for clinical management of HR-EBTs | Within 4 weeks after definitive surgical resection, prior to start of induction chemotherapy
  Feasibility of centralized diagnostics will be defined as:
  * 80% of patients will have central review and central molecular testing performed before timely start of therapy (~4 weeks post-surgery)
  Feasibility of national tumour board review will be defined as:
  * 80% of patients will be reviewed within treatment timeline of within ~4 weeks post-surgery
To establish a national HR infant brain tumor trial platform for future studies | At study completion (anticipated average duration of 2 years per participant)
  Data will be gathered on whether platform is able to support future research projects, facilitate collaboration in Canada, and improve clinical outcomes for this population

SECONDARY OUTCOMES:
To determine progression free and overall survival and patterns of failure for all enrolled patients | Up to 24 months following completion of maintenance therapy
  Time to progression (TTP), progression free survival (PFS) and overall survival (OS) up to two years following completion of treatment
To describe the toxicities of adding intrathecal (IT) chemotherapy and maintenance therapy after high dose chemotherapy for treatment of newly diagnosed HR-EBTs in patients less than 6 years of age | 30 days after last dose of study treatment
  Incidence of grade ≥3 adverse events (AE) and serious adverse events (SAE) related to study treatment

OTHER OUTCOMES:
To test the feasibility of prospective banking of tumor tissue, serial plasma and cerebrospinal fluid (CSF) for all enrolled patients | Through completion of study treatment (anticipated duration of 18-24 months per participant)
  To determine number of samples collected and bank CSF for potential future circulating tumour DNA (ctDNA analyses)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Cheng, Study Chair — BC Cancer Centre; Annie Huang, Study Chair — The Hospital for Sick Children; Lucie Lafay-Cousin, Study Chair — Alberta Children's Hospital
Locations (6):
- Canada (6):
  - Alberta Children's Hospital, Calgary, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - McMaster Children's Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
  - The Hospital for Sick Children, Toronto